CLINICAL TRIAL: NCT04377659
Title: A Phase II Study of IL-6 Receptor Antagonist Tocilizumab to Prevent Respiratory Failure and Death in Patients With Severe COVID-19 Infection
Brief Title: Tocilizumab for Prevention of Respiratory Failure in Patients With Severe COVID-19 Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on two large, multicenter, randomized trials showed no benefit to tocilizumab in this setting and study has been closed.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-185
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: COVD-19; Tocilizumab; Respiratory infection; 20-185; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intubation/Mechanical Ventilation (Experimental): Progression of respiratory failure in cohort #1 will be defined as a sustained increase in oxygen requirement or need for intubation/mechanical ventilation
  Interventions: Drug: Tocilizumab
- Respiratory Support (Experimental): In cohort #2 progression of respiratory failure will be defined as a need for increasing respiratory support (e.g. FiO2 or PEEP)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Participants will receive Tocilizumab 8 mg/kg i.v. at enrollment. Dose will be capped at 800 mg per infusion. If there is no improvement or toxicity, a second dose can be given 24 hrs to 5 days later.

SUMMARY:
The purpose of this study is to find out whether the study drug tocilizumab is an effective treatment for COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient or designated proxy willing and able to provide informed consent prior to enrollment in the study.
* COVID-19 PCR positive on nasopharyngeal swab
* Aged >/= 18 years old
* Patient hospitalized with newly diagnosed documented severe COVID-19 infection: with respiratory rate >/= 30 breaths/min OR peripheral capillary oxygen saturation (SpO2) < 93% on room air for nonintubated pts.
* Fever of 38.5 C or suspected respiratory infection
* IL-6 level >/= 80 pcg/ml
* Cohort #1 - non intubated Cohort #2 - intubated
* Women of childbearing potential must have a negative serum or urine pregnancy test
* Patients receiving ongoing steroid therapy are eligible
* Patients will be allowed to receive concurrent or sequential treatment with remdesivir

Exclusion Criteria:

* Patients with uncontrolled systemic fungal and bacterial infections
* Patients with latent tuberculosis
* Patients with known hypersensitivity to tocilizumab or any component of the formulation
* Concurrent initiation of steroid therapy is not allowed
* Patients with uncrontroled malignant disease, with a life expectancy of 3 months or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boglarka Gyurkocza, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intubation/Mechanical Ventilation | Respiratory Support
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intubation/Mechanical Ventilation | Respiratory Support | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Continuous [Median (Full Range); unit: years] | 68 [62 to 73] | 74 [64 to 87] | 73 [62 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression of Respiratory Failure or Death
Description: The primary endpoint for this cohort is progression of respiratory failure (binary yes/no while hospitalized). Progression of respiratory failure will be defined as a sustained increase in oxygen requirement (FiO2) or need for intubation/mechanical ventilation.
Time Frame: 14 days
Population: Data were not collected
Arm/Group | Intubation/Mechanical Ventilation | Respiratory Support
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intubation/Mechanical Ventilation | Respiratory Support
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intubation/Mechanical Ventilation (N=3) | Respiratory Support (N=6)
Thromboembolic Event (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
White Blood Cell Decreased (Investigations) | 0 | 1
Lymphocyte Count Decreased (Investigations) | 0 | 3
Infecions and Infestations - Other, specify - Covid-19 (Infections and infestations) | 0 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intubation/Mechanical Ventilation (N=3) | Respiratory Support (N=6)
Platelet count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 4
Anemia (Blood and lymphatic system disorders) | 3 | 2
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT04377659/Prot_SAP_000.pdf